CLINICAL TRIAL: NCT01910545
Title: PhaseI, Single-Center, Cohort Dose Escalation Trial to Determine the Safety, Tolerance, and Preliminary Antineoplastic Activity of OTS167, a MELK Inhibitor, in Patients With Refractory Locally Advanced or Metastatic Solid Tumor Malignancies
Brief Title: Phase 1 Study of OTS167 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoTherapy Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTS167-FR02
Record Dates: First submitted 2013-07-23; First posted 2013-07-29 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Solid Tumors; Metastatic Tumors
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OTS167IV (Experimental): single arm
  Interventions: Drug: OTS167IV

INTERVENTIONS:
Drug: OTS167IV

SUMMARY:
The purpose of this study is to test the safety and tolerability of an investigational drug called OTS167. OTS167 is a maternal embryonic leucine zipper kinase (MELK) inhibitor which demonstrated antitumor properties in laboratory tests. It is being developed as an anti-cancer drug. In this first-in-human study OTS167 will be administered to patients with solid tumors which have not responded to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, >= 18 years of age at the time of obtaining informed consent.
2. Patients with a documented (histologically- or cytologically-proven) solid tumor malignancy that is locally advanced or metastatic.
3. Patients with a malignancy that is either refractory to standard therapy or for which no standard therapy is available.
4. Patients with a malignancy that is currently not amenable to surgical intervention due to either medical contraindications or non-resectability of the tumor.
5. Patients with measurable or non-measurable disease according to the response evaluation criteria in solid tumors (RECIST , v1.1)
6. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
7. Patients, both male and female, who are either not of childbearing potential or who agree to use a medically effective method of contraception during the study and for 3 months after the last dose of study drug.
8. Patients with the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol.

Exclusion Criteria:

1. Women who are pregnant or lactating. Women of child-bearing potential (WOCBP), and fertile men with a WOCBP-partner not using adequate birth control.
2. Patients with known central nervous system (CNS) or leptomeningeal metastases not controlled by prior surgery or radiotherapy, or patients with symptoms suggesting CNS involvement for which treatment is required.
3. Patients with any hematologic malignancy. This includes leukemia (any form), lymphoma, and multiple myeloma.
4. Patients with any of the following hematologic abnormalities at baseline:

   * Absolute neutrophil count (ANC) < 1,500 per mm3
   * Platelet count < 100,000 per mm3
5. Patients with any of the following serum chemistry abnormalities at baseline:

   * Total bilirubin >= 1.5 × the ULN for the institution
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >= 3 × the upper limit normal (ULN) for the institution (>= 5 × if due to hepatic involvement by tumor)
   * Serum albumin < 2.5 g/dL
   * Creatinine >= 1.5 × ULN for the institution (or a calculated creatinine clearance < 60 mL/min/1.73 m2)
6. Patients with a significant cardiovascular disease or condition, including:

   * Congestive heart failure (CHF) currently requiring therapy
   * Need for antiarrhythmic medical therapy for a ventricular arrhythmia
   * Severe conduction disturbance
   * Angina pectoris requiring therapy
   * Corrected QT (QTc) interval > 450 msec (males) or > 470 msec (females)
   * QTc interval <= 300 msec
   * History of congenital long QT syndrome or congenital short QT syndrome
   * Left ventricular ejection fraction < 50%
   * Uncontrolled hypertension (per the Investigator's discretion)
   * Class III or IV cardiovascular disease according to the New York Heart Association's (NYHA) Functional Criteria.
   * Myocardial infarction (MI) within 6 months prior to first study drug administration
7. Patients with a known or suspected hypersensitivity to any of the components of OTS167.
8. Patients with a known history of human immunodeficiency virus (HIV) or active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV).
9. Patients with any other serious/active/uncontrolled infection, any infection requiring parenteral antibiotics, or unexplained fever > 38ºC within 1 week prior to first study drug administration.
10. Patients with inadequate recovery from acute toxicity associated with any prior antineoplastic therapy.
11. Patients with inadequate recovery from any prior surgical procedure, or patients having undergone any major surgical procedure within 4 weeks prior to first study drug administration.
12. Patients with any other life-threatening illness, significant organ system dysfunction, or clinically significant laboratory abnormality, which, in the opinion of the Investigator, would either compromise the patient's safety or interfere with evaluation of the safety of the study drug.
13. Patients with a psychiatric disorder or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary studies.
14. Patients with the inability or with foreseeable incapacity, in the opinion of the Investigator, to comply with the protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-08-23; Primary Completion 2016-04-11 (Actual); Study Completion 2016-05-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events and/or dose-limiting toxicities as a measure of safety and tolerability of OTS167 IV infusion. | Up to 30 days after last dose of study drug

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No